CLINICAL TRIAL: NCT07202312
Title: Clinical and Microbiological Efficacy of Ozone Therapy in the Non-surgical Treatment of Periodontal Disease
Brief Title: Ozone-therapy in Non-surgical Periodontal Therapy
Acronym: PD-OZONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alessia Pardo, PhD, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 698CET
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2023-08

CONDITIONS: Ozone-therapy (O3); Periodontitis; Antimicrobial Ozone Therapy
Keywords: ozone therapy; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone-therapy after non surgical therapy (Experimental): The test group received ozone therapy immediately after non-surgical treatment, at a fixed concentration of 2100 ppm and 80% oxygen, applied three times at the site. Ozone was delivered into the periodontal pocket using a sterile syringe with a flat tip. Ozone was generated with the Ozone DTA Ozone Generator (Denta Tec Dental AS, Norway), which was operated for 20 seconds in accordance with the manufacturer's instructions.
  Interventions: Device: Ozone-therapy after non-surgical therapy
- Non-surgical therapy (No Intervention): In the control group, non-surgical periodontal therapy was performed using both mechanical and manual instrumentation with curettes and ultrasonic devices.

INTERVENTIONS:
Device: Ozone-therapy after non-surgical therapy — The test group received ozone therapy immediately after non-surgical treatment, at a fixed concentration of 2100 ppm and 80% oxygen, applied three times at the site. Ozone was delivered into the periodontal pocket using a sterile syringe with a flat tip. Ozone was generated with the Ozone DTA Ozone Generator (Denta Tec Dental AS, Norway), which was operated for 20 seconds in accordance with the manufacturer's instructions.
  Arms: Ozone-therapy after non surgical therapy

SUMMARY:
Non-surgical periodontal therapy is a widely adopted procedure for the treatment of periodontitis, particularly in its moderate to severe stages. The approach involves the mechanical and manual debridement of subgingival biofilm and calculus through the use of ultrasonic scalers and hand curettes. This method aims to disrupt the pathogenic bacterial load within periodontal pockets and promote clinical attachment gain while reducing inflammation. However, the mechanical removal of biofilm alone may not always ensure complete bacterial eradication, especially in deep or anatomically complex sites.

To enhance bacterial disinfection and optimize clinical outcomes, the adjunctive use of ozone therapy has been introduced. This is a non-invasive technique that employs ozone in gaseous form to eliminate bacteria and fungi, inactivate viruses, and control bleeding. Its antiviral efficacy results from the denaturation of envelope proteins, impairment of viral adhesion to host cells, oxidation of unsaturated fatty acids within the lipid envelope, and degradation of single-stranded RNA. The synergistic effect of combining conventional non-surgical periodontal therapy with ozone therapy enables more thorough decontamination of periodontal pockets, even in cases where systemic antibiotics prove ineffective.

The aim of this study is to evaluate the clinical efficacy of adjunctive ozone therapy following non-surgical periodontal treatment in patients with severe periodontitis. The protocol consists of initial subgingival instrumentation using ultrasonic and manual tools, followed by the application of ozone therapy. The working hypothesis of this study is that the addition of ozone therapy provides superior bacterial reduction and improved clinical outcomes compared to mechanical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 84 years; Good general health status; Diagnosis of severe periodontitis involving at least 30% of all teeth, with at least three non-adjacent teeth presenting three sites with probing pocket depth (PPD) greater than 4 mm in at least two quadrants, and having lost at least four teeth due to periodontitis; Presence of at least 16 teeth, with a minimum of four teeth per quadrant.

Exclusion Criteria:

Pregnancy or breastfeeding; Presence of decompensated systemic diseases that may compromise the outcomes of the study or the patient's health; Regular use of antibiotics; Regular use of anti-inflammatory drugs (NSAIDs, corticosteroids, or aspirin); Use of anticoagulant medications; History of systemic antibiotic therapy within six months prior to enrollment; History of any periodontal therapy within six months prior to enrollment; Presence of severe mental or cognitive disorders.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth PPD Index | [Time Frame: T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (45 days after basline), T4 (3 months after baseline)]
  Probing depth is the distance from the gingival margin to the base of the pocket (mm)
Microbiological analysis | [Time Frame: T0 (Baseline), T2 (14 days after baseline), T3 (45 days after basline), T4 (3 months after baseline)]
  The microbiological analysis qualitatively (yes/no) assesses the presence of six types of periodontopathogenic bacteria (Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia, Treponema denticola, Actinomyces naeslundii) using sterile paper points inserted into the periodontal pocket prior to non-surgical periodontal therapy. For each site analyzed, two saliva samples are collected: one is placed in a test tube containing ethanol, and the other in a tube containing ammonium thioglycolate. The samples are subsequently transported to the microbiology department of the Integrated University Hospital of Verona for analysis.

SECONDARY OUTCOMES:
Recession REC Index | [Time Frame: T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (45 days after basline), T4 (3 months after baseline)]
  Recession is the apical shift of the marginal tissues associated with the attachment loss exposing the root or implant surface to the oral environment (mm)
Clinical attachment level CAL Index | [Time Frame: T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (45 days after basline), T4 (3 months after baseline)]
  measured in mm as distance from the CEJ to the gingival margin (GM)
Plaque Index | [Time Frame: T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (1 month after baseline), T4 (3 months after baseline)]
  This index ascertains the thickness of plaque along the gingival margin (%)
Bleeding on probing BOP Index | [Time Frame: T0 (Baseline), T1(7 days after baseline), T2 (14 days after baseline), T3 (1 month after baseline), T4 (3 months after baseline)]
  is an indicator of tissue inflammatory response to bacterial pathogens (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Alessia Pardo, Verona, Italy, Italy